## I1F-MC-RHCS Protocol b

A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects

NCT03848403

Approval Date: 30-May-2019

# Protocol I1F-MC-RHCS (b) A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects

## **Confidential Information**

The information contained in this protocol is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of ixekizumab (LY2439821), unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries.

**Note to Regulatory Authorities:** This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

Ixekizumab (LY2439821)

Eli Lilly and Company Indianapolis, Indiana USA 46285

Clinical Pharmacology Protocol Electronically Signed and Approved by Lilly: 29 October 2018.

Amendment (a) Electronically Signed and Approved by Lilly: 03 December 2018 Amendment (b) Electronically Signed and Approved by Lilly on date provided below.

Approval Date: 30-May-2019 GMT

# **Table of Contents**

# A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects

| Section | Page |
|---|---|
| Protocol I1F-MC-RHCS (b) A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects | 1 |
| Table of Contents | |
| 1. Protocol Synopsis | |
| 2. Schedule of Activities | |
| 3. Introduction | |
| 3.1. Study Rationale | |
| 3.2. Background | |
| 3.3. Benefit/Risk Assessment | |
| 4. Objectives and Endpoints | 19 |
| 5. Study Design. | |
| 5.1. Overall Design | |
| 5.2. Number of Participants | |
| 5.3. End of Study Definition | 21 |
| 5.4. Scientific Rationale for Study Design | 21 |
| 5.5. Justification for Dose | 21 |
| 6. Study Population | 23 |
| 6.1. Inclusion Criteria. | 23 |
| 6.2. Exclusion Criteria | 25 |
| 6.2.1. Rationale for Exclusion of Certain Study Candidates | 28 |
| 6.3. Lifestyle and/or Dietary Requirements | 28 |
| 6.3.1. Meals and Dietary Restrictions | |
| 6.3.2. Alcohol and Tobacco | 29 |
| 6.3.3. Activity | 29 |
| 6.4. Screen Failures | 29 |
| 7. Treatment | 30 |
| 7.1. Treatment Administered | 30 |
| 7.1.1 Packaging and Labeling | 31 |

| 7.2. Method of Treatment Assignment | 31 |
|-----------------------------------------------|---------------------|
| 7.2.1. Selection and Timing of Doses | 31 |
| 7.3. Blinding | 31 |
| 7.4. Dose Modification | 31 |
| 7.5. Preparation/Handling/Storage/Accountable | pility31 |
| 7.6. Treatment Compliance | 32 |
| 7.7. Concomitant Therapy | 32 |
| 7.8. Treatment after the End of the Study | 32 |
| 8. Discontinuation Criteria | 33 |
| 8.1. Discontinuation from Study Treatment | 33 |
| 8.1.1. Discontinuation of Inadvertently En | nrolled Subjects34 |
| 8.2. Discontinuation from the Study | 34 |
| 8.3. Subjects Lost to Follow-up | 34 |
| 9. Study Assessments and Procedures | 36 |
| 9.1. Efficacy Assessments | 36 |
| 9.2. Adverse Events | 36 |
| 9.2.1. Serious Adverse Events | 37 |
| 9.2.1.1. Adverse Events of Special Inter | est37 |
| 9.2.1.2. Suspected Unexpected Serious | Adverse Reactions38 |
| 9.2.2. Complaint Handling | 38 |
| 9.3. Treatment of Overdose | 39 |
| 9.4. Safety | 39 |
| 9.4.1. Laboratory Tests | 39 |
| 9.4.2. Vital Signs | 39 |
| 9.4.3. Electrocardiograms | 39 |
| 9.4.4. Temperature | 40 |
| 9.4.5. Other Tests | 40 |
| 9.4.5.1. Injection-Site Assessments | 40 |
| | 40 |
| 9.4.5.3. Injection-Site Pain | 40 |
| - | ng Scale41 |
| 1 2 1 | rale41 |
| | 41 |
| 1 | 41 |
| | 42 |
| | 42 |
| _ · | 42 |
| 0.7 Genetics | 42 |

| I1F-MC-RHCS Clinical Pharmacology Protocol (b) | Page 4 |
|---------------------------------------------------------------|--------|
| 9.8. Biomarkers | 43 |
| 9.9. Health Economics | 43 |
| 10. Statistical Considerations and Data Analysis | 44 |
| 10.1. Sample Size Determination | |
| 10.2. Populations for Analyses | 44 |
| 10.2.1. Study Participant Disposition | 44 |
| 10.2.2. Study Participant Characteristics | 44 |
| 10.3. Statistical Analyses | 44 |
| 10.3.1. Safety Analyses | 45 |
| 10.3.1.1. Clinical Evaluation of Safety | 45 |
| 10.3.1.2. Statistical Evaluation of Safety | 45 |
| 10.3.1.2.1. Injection-Site Pain | 45 |
| 10.3.1.2.2. Statistical Evaluation of Other Safety Parameters | 45 |
| 10.3.2. Data Review During the Study | 45 |
| 10.3.3. Interim Analyses | 46 |
| 11. References | 47 |

| 11F-MC-RHCS | Clinical | Pharmacolog | qv | Protocol ( | (b) |
|-------------|----------|-------------|----|------------|-----|
|-------------|----------|-------------|----|------------|-----|

| Ρ | aç | 1e | 5 |
|---|----|----|---|

# **List of Tables**

| Table | | Page |
|---------------|--------------------------|------|
| Table RHCS.1. | Objectives and Endpoints | 19 |
| Table RHCS.2. | Treatments Administered | 30 |

| 11F-MC-RHCS C | linical Pharmacology Protocol (b) | Page 6 |
|---|---|---|
| | List of Figures | |
| Figure | | Page |
| Figure RHCS.1. | Illustration of study design for Protocol I1F-MC-RHCS | 21 |

# **List of Appendices**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Abbreviations and Definitions | 48 |
| Appendix 2. | Clinical Laboratory Tests | 52 |
| Appendix 3. | Study Governance, Regulatory and Ethical Considerations | 54 |
| Appendix 4. | Hepatic Monitoring Tests for Treatment-Emergent Abnormality | 57 |
| Appendix 5. | Blood Sampling Summary | 58 |
| Appendix 6. | Protocol Amendment I1F-MC-RHCS (b) Summary: A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects | 59 |
| | Syringe in Healthy Subjects | 39 |

# 1. Protocol Synopsis

#### Title of Study:

A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects

#### Rationale:

Changes in buffer composition are being investigated as a potential way to address injection-site pain reported for ixekizumab. Study I1F-MC-RHCS is therefore being conducted to compare injection-site pain and tolerability of ixekizumab administered using 2 new formulations, compared to the commercial formulation.

#### **Objective/Endpoint:**

| Objective | Endpoint |
|---|---|
| Primary | |
| Evaluate pain intensity on injection of ixekizumab with different formulations. | Visual analog scale (VAS) pain score immediately (within 1 minute) after injection |

#### **Summary of Study Design:**

This will be a single-dose, subject-blind, 3-period, 3-treatment, randomized, crossover study in healthy subjects. Eligible subjects will be admitted to the clinical research unit (CRU) on Day -1 and randomized 1:1:1 to 1 of 3 possible treatment sequences.

Subjects may be allowed to leave the CRU after completing the 4-hour safety assessments for Day 1, at the investigator's discretion. Subjects will be readmitted to the CRU on Days 7 and 14 to receive their second and third injections on Days 8 and 15, respectively, and may be allowed to leave the CRU after completing the 4-hour safety assessments at the investigators discretion on Days 8 and 15, respectively. Subjects will return to the CRU as an outpatient on Days 21 ( $\pm 1$  day) and 43 ( $\pm 3$  days) for a safety check-up. In addition, safety follow-up telephone calls will be conducted in between outpatient visits, on Days 28 ( $\pm 1$  day), 35 ( $\pm 3$  days), 50 ( $\pm 3$  days), 57 ( $\pm 3$  days), and 64 ( $\pm 3$  days), with a final safety follow-up telephone call on Day 71 ( $\pm 3$  days). There will be a follow-up visit approximately 12 weeks after the last injection.

Safety and tolerability will be assessed by monitoring of adverse events (AEs), injection-site assessments, injection-site pain, bleeding/bruising assessments, Columbia Suicide Severity Rating Scale (C-SSRS), Hospital Anxiety Depression Scale (HADS), vital signs assessments, temperature, physical examination, 12-lead electrocardiograms (ECGs), and clinical laboratory tests. Pain assessments will be made using an injection-site visual analog scale (VAS).

#### Treatment Arms and Planned Duration for an Individual Subject:

All subjects will be screened within 28 days prior to enrollment. On Days 1, 8, and 15, subjects will receive a single 1-mL subcutaneous injection of 1 of the following treatments, according to the randomization schedule:

• 80 mg ixekizumab Commercial Formulation (Reference)

- 80 mg ixekizumab Test Formulation 1
- 80 mg ixekizumab Test Formulation 2

Subjects will participate in the study for approximately 18 weeks.

#### **Number of Subjects:**

Up to 102 subjects may be enrolled to maximize the intent to have 78 subjects (26 in each treatment sequence) complete the study. Attempts will be made to enroll a total of 3 Japanese completers.

#### **Statistical Analysis:**

Abnormal lab values will be listed. Other safety parameters that will be assessed include injection-site assessments, including pain, induration, swelling, pruritus, bleeding/bruising, and erythema/redness. The parameters will be listed, and summarized using standard descriptive statistics. Suicidal ideation and/or behavior and self-injurious behavior with no suicidal intent, based on the C-SSRS, will be listed by subject. HADS item scores will be listed for subjects with HADS depression subscale  $\geq 11$  at any time. Additional analyses may be performed if warranted upon review of the data.

VAS pain score will be summarized using standard descriptive statistics. In addition, the severity of pain will be categorized by VAS pain score as: mild pain ( $\leq$ 30), moderate pain (>30 and  $\leq$ 70), and severe pain (>70). The number and percentage of the subjects in each pain severity category will be summarized by treatment and time point.

# 2. Schedule of Activities

**Study Schedule Protocol I1F-MC-RHCS** 

| Study Schedu | Screening | - | Study Day | | | | | | | | | | | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days 50, 57, & 64 (± 3 days) | Day 71 (± 3 days) | | |
| Informed<br>Consent | X | | | | | | | | | | | | | |
| Subject<br>Admission to<br>CRU | | X | | X | | X | | | | | | | | |
| Subject Discharge from CRU | | | X | | X | | X | | | | | | | |
| Safety<br>Assessment<br>(Telephone<br>Call) | | | | | | | | | X | | X | X | | Every effort will be made to contact subjects as near to this time as possible but missed calls will not be recorded as protocol deviations. |
| Medical History<br>and<br>Demographics | X | | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | |
| Weight | X | X | | | | | | | | | | | X | |
| Serology | X | | | | | | | | | | | | | |
| QuantiFERON® -TB Gold or TST | X | | | | | | | | | | | | | |
| Randomization | | | X | | | | | | | | | | | |

| | Screening | | | | | | Study Da | ay | | | | | FU/<br>ED <sup>a</sup> | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days<br>50,<br>57, &<br>64<br>(± 3<br>days) | Day 71 (± 3 days) | | |
| Investigational<br>Product<br>Administration | | | X | | X | | X | | | | | | | |
| Ethanol Testing<br>and Urine Drug<br>Screen | X | X | | X | | X | | | | | | | | May be repeated at the discretion of the investigator. |
| Pregnancy Test<br>(Females Only;<br>as applicable) | X | X | | X | | X | | | | | | | X | Serum pregnancy test will be performed at screening. Urine pregnancy test will be performed at all subsequent time points. |
| FSH Test | X | | | | | | | | | | | | | Females only, if applicable. |
| Physical Exam | | X | | | | | | | | | | | X | After baseline exam,<br>medical assessment is<br>performed only to include<br>medical review and<br>targeted examination, as<br>appropriate. |
| 12-lead ECG | X | | | | | | | | | | | | X | Single readings will be taken after at least 5 minutes in a supine position. |

| | Screening | | Study Day | | | | | | | | | | | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days 50, 57, & 64 (± 3 days) | Day 71 (± 3 days) | | |
| HADS<br>Depression<br>sub-scale | X | X | | X | | X | | X | | X | | | X | |
| C-SSRS and<br>Lilly Self-Harm<br>Supplement | Х | X | | X | | X | | X | | X | | | X | At screening 'Baseline -<br>Screening' questionnaire<br>to be used, all other<br>timepoints use 'Since Last<br>Visit' questionnaire. |
| Body<br>Temperature | | | P | X | | X | | X | | X | | | X | |
| Clinical<br>Chemistry,<br>Hematology,<br>and Urinalysis<br>Tests | Х | X | | X | | X | | X | | X | | | X | See Appendix 2, Clinical<br>Laboratory Tests, for<br>details. |

| | Screening | Study Day | | | | | | | | | | FU/<br>ED <sup>a</sup> | Comments | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days 50, 57, & 64 (± 3 days) | Day 71 (± 3 days) | | |
| Injection-Site<br>Assessments<br>(Minutes) | | | 0, 10,<br>20,<br>30,<br>60,<br>120,<br>240 | | 0,<br>10,<br>20,<br>30,<br>60,<br>120,<br>240 | | 0, 10,<br>20,<br>30,<br>60,<br>120,<br>240 | X | | X | | | | Assessments of induration, swelling, pruritus, and erythema/redness (collected as described in Section 9.4.5.1). 0-minute time point should be done within 1 minute following injection; within ± 2 minutes of the 10, 20, and 30-minute time points; within ± 5 minutes of the 60, 120, and 240-minute time points. Assessments will be conducted once during the 1-week follow-up on Day 21 (± 1 day) and on Day 43 (± 3 days). |
| Injection-Site Pain Assessment using VAS (Minutes) | | | 0, 10,<br>20,<br>30, 60 | | 0,<br>10,<br>20,<br>30,<br>60 | | 0, 10,<br>20,<br>30, 60 | | | | | | | Assessment of injection-site pain (VAS) at the 0-minute time point should be done within 1 minute following injection; within $\pm$ 2 minutes of the 10, 20, and 30-minute time points; within $\pm$ 5 minutes of the 60-minute time point. |
| | Screening | 5 | | Study Day | | | | | | | | | FU/<br>ED <sup>a</sup> | Comments |

| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days<br>50,<br>57, &<br>64<br>(±3<br>days) | Day 71 (± 3 days) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Injection-Site Bleeding/Bruising Assessment (Minutes) | | | 0,<br>10,<br>20,<br>30,<br>60,<br>120,<br>240 | | 0,<br>10,<br>20,<br>30,<br>60,<br>120,<br>240 | | 0, 10,<br>20,<br>30,<br>60,<br>120,<br>240 | X | | X | | | | Observational assessment of injection-site bleeding and bruising. 0-minute time point should be done within 1 minute following injection; within ± 2 minutes of the 10, 20, and 30-minute time points; within ± 5 minutes of the 60, 120, and 240-minute time points. |
| Pharmacokinetic<br>Sample | | | | | | | | X | | | | | X | Samples to be stored only. |
| Immunogenicity<br>Sample | | X | | | | | | X | | | | | X | Samples to be stored only. |
| Vital Signs<br>(Sitting) | X | X | P,<br>2-4 | Х | P,<br>2-4 | Х | P, 2-4 | X | | X | | | Х | Day 1, 8, and 15: 2-4 hour assessment to be conducted at least 2 hours postdose and prior to discharge at approximately 4 hours postdose. Sitting blood pressure and pulse rate may be measured as clinically indicated. Timepoints may be added if warranted. |

| | Screening | | | | Study Day | | | | | | | | FU/<br>ED <sup>a</sup> | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2<br>days prior<br>to Day 1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day 21 (± 1 day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day<br>43<br>(± 3<br>days) | Days 50, 57, & 64 (± 3 days) | Day 71 (± 3 days) | | |
| Pharmacogenetic Sample | | X | | | | | | | | | | | | |
| Adverse Events<br>and Concomitant<br>Medication | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Abbreviations: CRU = clinical research unit; C-SSRS = Columbia Suicide Severity Rating Scale; ECG = electrocardiogram; ED = early discontinuation; FSH = follicle-stimulating hormone; FU = follow-up; HADS = Hospital Anxiety and Depression Scale; P = predose; TB = tuberculosis; TST = tuberculin skin test; VAS = visual analog scale.

Note: if multiple procedures take place at the same time point, the following order should be used: ECG, vital signs, and venipuncture.

<sup>&</sup>lt;sup>a</sup> Follow-up / Early Discontinuation should be  $\sim$ 12 weeks post last injection ( $\pm$ 1 week).

## 3. Introduction

## 3.1. Study Rationale

Ixekizumab is administered subcutaneously (SC), and is available as an injectable solution in either a manual prefilled syringe (PFS) or a 1-mL autoinjector (AI).

Study I1F-MC-RHCK was conducted to assess acute pain and injection site reactions following administration of ixekizumab via marketed AI (fast injection speed, visible needle), a modified AI (slow injection speed, hidden needle), the marketed PFS, and placebo administered using a device similar to the marketed AI (fast injection speed, visible needle). The results showed no statistically significant difference in intensity of injection-site pain following single injections administered via any of the methods tested. Safety profiles, including frequency of injection site reactions (ISRs), were also similar between treatments.

Several solution-associated factors may contribute to pain perception associated with injectable therapeutics, including active pharmaceutical ingredient, pH, buffer composition, and tonicity (Laursen et al. 2006).

Two new formulations of ixekizumab have therefore been developed using alternative approaches for buffer and tonicity agent. Neither have been tested in humans or animals thus far.



Study RHCS is being conducted in parallel with Study I1F-MC-RHCT which will provide further assessment of the pharmacokinetics of ixekizumab and injection-site pain and ISRs associated with administration of the 3 ixekizumab formulations in a parallel-design study.

# 3.2. Background

Ixekizumab (LY2439821, Taltz®) is a humanized immunoglobulin G subclass 4 monoclonal antibody that binds with high affinity and specificity to interleukin (IL)-17A, a proinflammatory cytokine. Ixekizumab is marketed in the US and EU for the treatment of moderate-to-severe psoriasis (Ps) at a dose of 160 mg at Week 0, followed by 80 mg every 2 weeks (Q2W) up to Week 12, then maintenance dosing of 80 mg every 4 weeks (Q4W), and for active psoriatic arthritis at a dose of 160 mg at Week 0 followed by 80 mg Q4W. In Japan, ixekizumab is marketed for moderate-to-severe plaque Ps, erythrodermic Ps, pustular Ps, and psoriatic arthritis.

#### 3.3. Benefit/Risk Assessment

As this study will enroll healthy subjects, there is no anticipated therapeutic benefit for the subjects.

As of the cut-off date for the current Investigator's Brochure (IB; 22 March 2018), more than 8755 clinical trial subjects have received at least 1 dose of ixekizumab (5934 patients with Ps,

532 patients with rheumatoid arthritis, 1301 patients with psoriatic arthritis, 119 healthy subjects, and an estimated 869 patients with axial spondyloarthritis).

Forty-one healthy subjects were administered ixekizumab by PFS (160 mg [2 × 80 mg] followed by 80 mg 2 weeks later) in Study I1F-MC-RHCA (Study RHCA). All adverse events (AEs) in Study RHCA were mild in severity. The most commonly reported AEs were headache, injection-site erythema, and fatigue. With the exception of fatigue, this is consistent with commonly reported AEs reported in Phase 3 trials. An additional 78 healthy subjects were administered ixekizumab by PFS, marketed AI, and modified AI (3 single 80 mg doses) in Study I1F-MC-RHCK. All treatment-emergent AEs (TEAEs) were mild in severity and the most commonly reported TEAEs were ISRs, injection site pruritus, nausea, diarrhea, upper respiratory tract infection, and injection-site erythema. Pharmacokinetic simulations (described further in Section 5.5) show that the 80 mg dose given every week for a total of 3 injections proposed for this study is projected to give exposures that are within the range of exposure to ixekizumab reported in previous studies, thus a similar TEAE profile is expected. The excipients are expected to be safe and well tolerated.

More information about the known and expected benefits, risks, serious AEs (SAEs) and reasonably anticipated AEs of ixekizumab are to be found in the IB.

# 4. Objectives and Endpoints

Table RHCS.1 shows the objectives and endpoints of the study.

# Table RHCS.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| <u>Primary</u> | |
| Evaluate pain intensity on injection of ixekizumab with | Visual analog scale (VAS) pain score immediately |
| different formulations. | (within 1 minute) after injection |
| Exploratory | |
| To evaluate the safety and tolerability of a single 80 mg | TEAEs, SAEs, ISRs, and VAS pain scores |
| SC dose of ixekizumab Test Formulation 1 and Test | |
| Formulation 2 formulations compared to the commercial | |
| formulation (Reference) | |

# 5. Study Design

# 5.1. Overall Design

This will be a single-dose, subject-blind, 3-period, 3-treatment, randomized, crossover study in healthy subjects.

All subjects will be screened within 28 days prior to enrollment. Eligible subjects will be admitted to the clinical research unit (CRU) on Day -1 and randomized 1:1:1 to 1 of 3 possible treatment sequences (see Figure RHCS.1). On Day 1, subjects will receive a single 1-mL SC injection of 1 of the following treatments, according to the randomization schedule:

- 80 mg ixekizumab Commercial Formulation (Reference)
- 80 mg ixekizumab Test Formulation 1
- 80 mg ixekizumab Test Formulation 2

Subjects may be allowed to leave the CRU after completing the 4-hour safety assessments for Day 1, at the investigator's discretion. Subjects will be readmitted to the CRU on Days 7 and 14 to receive their second and third injections on Days 8 and 15, respectively, and may be allowed to leave the CRU after completing the 4-hour safety assessments at the investigators discretion on Days 8 and 15, respectively. Subjects will return to the CRU as an outpatient on Days 21 ( $\pm$  1 day) and 43 ( $\pm$  3 days) for a safety check-up. In addition, safety follow-up telephone calls will be conducted in between outpatient visits, on Days 28 ( $\pm$  1 day), 35 ( $\pm$  3 days), 50 ( $\pm$  3 days), 57 ( $\pm$  3 days), and 64 ( $\pm$  3 days), with a final safety follow-up telephone call on Day 71 ( $\pm$  3 days). There will be a follow-up visit approximately 12 weeks after the last injection.

Site staff will administer all injections. All injections will be administered in the abdomen while the subject is in a sitting or a reclining position. Subsequent injections will be alternated between the abdominal quadrants. The injection site will be documented. Injections should not be made into an area that shows evidence of bruising, redness, or a rash from a previous injection. All study injection sites will be marked for size and with a surgical marker in order to identify study injection sites. Every attempt will be made to have injections for individual subjects be performed by the same clinical staff member.

Injection-site assessments will be administered immediately after each injection and at 10, 20, 30, 60, 120, and 240 minutes post injection. The injection-site pain VAS will be administered immediately after each injection and at 10, 20, 30, and 60 minutes post-injection.

Safety and tolerability will be assessed by monitoring of AEs, injection-site assessments, injection-site pain, bleeding/bruising assessments, Columbia Suicide Severity Rating Scale (C-SSRS), Hospital Anxiety and Depression Scale (HADS), vital signs assessments, temperature, physical examination, 12-lead electrocardiograms (ECGs), and clinical laboratory tests.

Study governance considerations are described in detail in Appendix 3.

Figure RHCS.1 illustrates the study design.

#### Group 1



Subjects will be blinded to all treatments.

Figure RHCS.1. Illustration of study design for Protocol I1F-MC-RHCS.

## 5.2. Number of Participants

Up to 102 subjects may be enrolled to maximize the intent to have 78 subjects (26 subjects per treatment sequence) complete the study. For purposes of this study, a subject completes the study when all procedures scheduled for Day 21 have been finished. Attempts will be made to enroll a total of 3 Japanese completers.

# 5.3. End of Study Definition

End of the study is the date of the last visit or last scheduled procedure shown in the Schedule of Activities (Section 2) for the last subject.

# 5.4. Scientific Rationale for Study Design

Healthy subjects have been chosen for this exploratory study so that potential formulations may be explored prior to conducting trials in target patient populations.

The study has a 3-period crossover design to allow each subject to act as their own control. This design allows a comparison of the effects of ixekizumab administered using the commercial formulation to Test Formulation 1 and Test Formulation 2. All injections will be administered in the abdomen for consistency, because the abdomen is one of the most commonly used sites for self-injection in clinical practice.

#### 5.5. Justification for Dose

The recommended dose for Ps patients is 160 mg by SC injection (two 80-mg injections) at Week 0, followed by an 80-mg injection at Weeks 2, 4, 6, 8, 10, and 12, then 80 mg Q4W. The

dosing regimen in Study RHCS is not designed to mimic that used in clinical practice but to administer the commercial dose strength (80 mg/mL), since the primary objective is evaluation of the pain that occurs within 1 hour of the time of injection. Subjects in Study RHCS will receive a total of 3 injections of 80 mg ixekizumab separated by 1-week intervals (total dose 240 mg).

Across studies in Ps patients, doses of ixekizumab from 5 to 160 mg SC and 15 mg intravenously have been studied, given on a Q2W or Q4W basis. In addition, studies in rheumatoid arthritis patients evaluated doses up to 180 mg Q2W and 120 mg weekly. Pharmacokinetic simulations of the ixekizumab dose regimens proposed for Study RHCS were compared to pharmacokinetic data in healthy subjects in Study RHCA and in patients with Ps. These pharmacokinetic simulations show that the 80 mg dose given every week for a total of 3 injections proposed for this study is projected to give exposures that are within the range of exposure to ixekizumab reported in previous studies, thus a similar TEAE profile is expected (see Section 3.3).

# 6. Study Population

Eligibility of subjects for the study will be based on the results of medical history, vital signs, clinical laboratory tests, electrocardiogram (ECG), and physical examination.

The nature of any conditions present at the time of the physical examination and any preexisting conditions will be documented. Screening and/or Day -1 laboratory testing may be repeated once at the discretion of the investigator for any out of range results.

Screening may occur up to 28 days prior to enrollment. Subjects who are not enrolled within 28 days of screening may be subjected to an additional medical assessment and/or clinical measurements to confirm their eligibility.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, are not permitted.

#### 6.1. Inclusion Criteria

Subjects are eligible for inclusion in the study only if they meet all of the following criteria at screening and/or Day -1:

[1] are overtly healthy males or females, as determined by screening medical history and physical examination, or are males or females with chronic, stable medical problems that, in the investigator's opinion, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.

#### [1a] male subjects:

agree to use a reliable method of birth control and to not donate sperm during the study and for 3 months following the last dose of ixekizumab.

Examples of reliable methods of birth control are condoms with spermicide, oral contraceptives or intrauterine device used by the female partner, and male sterilization

Subjects who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either maintain abstinence or stay in a same-sex relationship without sexual relationships with females. Periodic abstinence, declaration of abstinence just for the duration of the trial, and withdrawal are not acceptable methods of contraception.

#### [1b] female subjects:

1) must be women of child-bearing potential who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either remain abstinent or stay in a same-sex relationship without sexual relationships with males. Periodic abstinence (eg, calendar, ovulation, symptothermal,

- post-ovulation methods), declaration of abstinence just for the duration of the trial, and withdrawal are not acceptable methods of contraception.
- 2) Otherwise, women of child-bearing potential must agree to use 1 highly effective method (less than 1% failure rate) of contraception, or a combination of 2 effective methods of contraception for the entirety of the study and for 3 months following the last dose of ixekizumab.
  - i. Women of child-bearing potential participating must test negative for pregnancy prior to initiation of treatment as indicated by a negative serum pregnancy test at the screening visit followed by a negative urine pregnancy test within 24 hours prior to exposure to study drug at each entry to the CRU.
  - ii. Either 1 highly-effective method of contraception (such as combination oral contraceptives, implanted contraceptives, or intrauterine device) or a combination of 2 effective methods (such as male or female condoms with spermicide, diaphragms with spermicide, or cervical sponges) will be used. The subject may choose to use a double-barrier method of contraception. Barrier protection methods without concomitant use of a spermicide are not a reliable or acceptable method. Thus, each barrier method must include use of a spermicide. It should be noted that the use of male and female condoms as a double-barrier method is not considered acceptable due to the high failure rate when these methods are combined.
- 3) Women not of child-bearing potential may participate and include those who are:
  - i. infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation, or permanent tubal occlusion such as Essure), a congenital anomaly such as mullerian agenesis; or
  - ii. post-menopausal defined as either:
    - a) a woman at least 50 years of age with an intact uterus, not on hormone therapy, who has had either:
      - cessation of menses for at least 1 year; or
      - at least 6 months of spontaneous amenorrhea with a follicle-stimulating hormone level >40 mIU/mL.
    - b) a woman 55 years or older, not on hormone therapy, who has had at least 6 months of spontaneous amenorrhea;

- c) a woman 55 years or older with a diagnosis of menopause prior to starting hormone replacement therapy.
- [2] are aged at least 18 (20 for Japanese subjects) to 75 years at the time of screening.
- [3] have a body mass index (BMI) of 18.0 to 32.0 kg/m<sup>2</sup>, inclusive at screening.
- [4] have venous access sufficient to allow for blood sampling as per the protocol.
- [5] are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
- [6] are able and willing to give informed consent.
- [7] For Japanese subjects, the subject, the subject's biological parents, and all of the subject's biological grandparents must be of exclusive Japanese descent and born in Japan.

#### 6.2. Exclusion Criteria

Subjects will be excluded from study enrollment if they meet any of the following criteria at screening and/or Day -1:

- [8] are investigative site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, biological or legal guardian, child, or sibling.
- [9] are Lilly, or Covance employees.
- [10] are currently enrolled in a clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study.
- [11] have participated, within the last 30 days, in a clinical study involving an IP. If the previous IP has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed.
- [12] have previously completed or withdrawn from this study or any other study investigating ixekizumab, and have previously received ixekizumab, or have ever been administered other IL-17 antagonists.
- [13] have known allergies to ixekizumab, related compounds or any components of the formulations, or history of significant atopy.
- [14] have self-perceived dullness or loss of sensation on either side of their abdomen.
- [15] have uncontrolled arterial hypertension characterized by a systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg.
  - Note: if an initial blood pressure reading exceeds this limit, the reading may be repeated once after the subject has rested sitting for  $\geq 10$  minutes. If the repeat value is less than the criterion limits, the second value may be accepted.

- [16] have a significant history of, or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or hematologic disorders, that in the opinion of the investigator poses an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of data.
- [17] Presence of significant uncontrolled neuropsychiatric disorder; have lifetime history of suicidal behavior (yes to any suicidal behavior question from the "Suicidal Behavior" portion of the C-SSRS from screening and between screening and baseline [Day -1]); have history of active suicidal ideation within the past year (yes to question 4 or 5 on the "Suicidal Ideation" portion of the C-SSRS from screening and between screening and baseline [Day-1]) and/or are clinically judged by the investigator to be at risk for suicide.
- [18] Have recent history (past 30 days) of depression; have HADS Depression subscale score of >11.
- [19] Have current or history of inflammatory bowel disease (IBD) (Crohn's disease or ulcerative colitis), or signs or symptoms indicative of ulcerative colitis or Crohn's disease (based on investigator determination), or knowledge of a family history of IBD in first degree relatives.

#### [20] Infections:

[20a] have had a serious infection (e.g., pneumonia, cellulitis, and sepsis), have been hospitalized, or have received intravenous antibiotics for an infection within 12 weeks prior to Day 1; have had a serious bone or joint infection within 24 weeks prior to Day 1, or have ever had an infection of an artificial joint; or are immunocompromised to an extent such that participation in the study would post an unacceptable risk to the subject.

[20b] Have or have had an infection typical of an immunocompromised host and/or that occurs with increased incidence in an immunocompromised host (including, but not limited to, pneumocystis jiroveci pneumonia, histoplasmosis, or coccidioidomycosis), or have a known immunodeficiency.

[20c] Have or have had a herpes zoster infection or any other clinically apparent varicella-zoster virus infection within 12 weeks of Day 1.

[20d] Have had any other active or recent infection within 4 weeks of Day 1 that, in the opinion of the investigator would pose an unacceptable risk to the subject if participating in the study; these subjects may be re-screened (once)  $\geq$ 4 weeks after documented resolution of symptoms.

- [21] have a history of uncompensated heart failure, fluid overload, or myocardial infarction, or evidence of new-onset ischemic heart disease or other serious cardiac disease, within 12 weeks prior to Day 1.
- [22] have clinical laboratory test results at screening that are outside the normal reference range for the population and are considered clinically significant, and/or have any of the following specific abnormalities:

- neutrophil count <1500 cells/μL
- lymphocyte count <800 cells/μL
- platelet count <100,000 cells/μL
- total white blood cell count <3000 cells/μL

Note: laboratory tests may be repeated if there is a documented technical error, or once at the discretion of the investigator for any out of range results.

- [23] regularly use known drugs of abuse and/or show positive findings on drug screening.
- [24] show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies.
- [25] show evidence of hepatitis C and/or positive hepatitis C antibody.
- [26] show evidence of, or test positive for hepatitis B and/or positive hepatitis B surface antigen and/or hepatitis B core antibody.
- [27] are women who are lactating.
- [28] have donated blood of more than 500 mL within the last month prior to dosing or intend to donate blood during the course of the study.
- [29] have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (females up to and over 65, and males over 65), or are unwilling to stop alcohol consumption for 48 hours prior to each admission to the CRU until CRU discharge, plus 48 hours prior to admission to the CRU for the 12-week follow-up visit until final discharge from the CRU, or are unwilling to restrict alcohol intake to 3 units per day (males) and 2 units per day (females) between CRU admission periods (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
- [30] show evidence of active or latent tuberculosis (TB), as documented by medical history and examination, any recent chest x-rays (if obtained in the previous 6 months; x-rays will not be taken for the sole purpose of determining eligibility for this study), and TB testing: either a positive tuberculin skin test (TST; defined as a skin induration >5 mm at 48 to 72 hours, regardless of Bacillus Calmette-Guérin [BCG] or other vaccination history), or a positive (not indeterminate) QuantiFERON®-TB Gold test. The choice to perform a TST or a QuantiFERON-TB Gold test will be made by the investigator according to local licensing and standard of care. The QuantiFERON-TB Gold test can only be used in countries where it is licensed, and the use of this test is dependent on previous treatment(s). This test may not be suitable if previous treatment(s) produce significant immunosuppression.

[31] had a vaccination with BCG, other live vaccines, or attenuated live vaccines within 12 months prior to first admission to the CRU, or intend to have a vaccination with BCG during the course of the study, or within 12 months of completing treatment in this study.

Note: killed/inactive or subunit vaccines are expected to be safe; however, their efficacy with concomitant ixekizumab is unknown.

- [32] have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
- [33] intend or are likely to use over-the-counter or prescription medication for pain or inflammation within 7 days prior to each dose administration. Subjects on stable doses of other medications (for example, statins and anti-hypertensives) may be eligible for enrollment following discussion with the Sponsor (Section 7.7).
- [34] have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the subject if participating in this study.
- [35] have had any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
- [36] have any condition that could affect pain perception from an injection.
- [37] have excessive tattoos or scars over the abdomen, or other factors (eg, rash, excessive folds of skin) that, in the investigator's opinion, would interfere with injection-site assessments.
- [38] in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.

# 6.2.1. Rationale for Exclusion of Certain Study Candidates

Exclusion criteria [8] and [9] prevent conflict of interest in study participants. Exclusion criteria [10] through [38] exclude items including, but not limited to, medical conditions, medication intolerance, and concomitant medication use that may confound the assessment of study endpoints.

# 6.3. Lifestyle and/or Dietary Requirements

Throughout the study, subjects may undergo medical assessments and review of compliance with requirements before continuing in the study. Subjects will also be required to adhere to contraceptive requirements, as outlined in the inclusion criteria (Section 6.1).

# 6.3.1. Meals and Dietary Restrictions

Subjects will receive a light breakfast on the morning of Days 1, 8, and 15, but will be fasted (water is permitted) from 1 hour prior to dosing until 1 hour postdose. Standard meals will be provided at all other times while subjects are resident at the CRU, per the CRU's policy.

#### 6.3.2. Alcohol and Tobacco

Subjects should not drink alcohol for 48 hours prior to each admission to the CRU until CRU discharge, plus 48 hours prior to admission to the CRU for the 12-week follow-up visit until final discharge from the CRU. Alcohol intake between CRU admission periods should not exceed 3 units per day (males) and 2 units per day (females). In addition, subjects must abide by the CRU smoking restrictions during study visits and whilst resident in the CRU.

## 6.3.3. Activity

Subjects will be encouraged to maintain their regular exercise; however, they should not undertake vigorous or prolonged exercise within 48 hours prior to each CRU visit.

#### 6.4. Screen Failures

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened once at the investigator's discretion (see Section 6).

## 7. Treatment

#### 7.1. Treatment Administered

A dose of IP will consist of 1 SC injection of 80 mg ixekizumab into the abdomen. All doses will be administered by clinical site staff.

The study involves a comparison of:

- 80 mg ixekizumab Commercial Formulation administered SC via PFS (Reference)
- 80 mg ixekizumab Test Formulation 1 administered SC via PFS (Test Formulation 1)
- 80 mg ixekizumab Test Formulation 2 administered SC via PFS (Test Formulation 2)

Prior to the PFS injection, the investigator or his/her designee will clean the subject's skin. The injection will be administered by clinical site staff, according to the instructions provided by the sponsor.

Table RHCS.2 shows the treatment regimens.

Table RHCS.2. Treatments Administered

| Treatment Name | Reference | Test Formulation 1 | Test Formulation 2 |
|---|---|---|---|
| Formulation | solution for injection | solution for injection | solution for injection |
| Dose | 80 mg ixekizumab | 80 mg ixekizumab | 80 mg ixekizumab |
| Route of Administration | SC injection | SC injection | SC injection |
| <b>Delivery Method</b> | PFS | PFS | PFS |

Abbreviations: PFS = prefilled syringe; SC = subcutaneous.

The investigator or designee is responsible for:

- explaining the correct use of the IPs to the site personnel
- verifying that instructions are followed properly
- maintaining accurate records of IP dispensing and collection
- and returning all unused medication to Lilly or its designee at the end of the study

**Note:** In some cases, sites may destroy the material if, during the investigative site selection, the evaluator has verified and documented that the site has appropriate facilities and written procedures to dispose of clinical materials.

## 7.1.1. Packaging and Labeling

Ixekizumab will be supplied by the sponsor or its designee in accordance with current good manufacturing practice, labeled according to the country's regulatory requirements, and supplied with lot numbers, expiry dates, and certificates of analysis, as applicable.

Each syringe of ixekizumab is designed to deliver 80 mg of ixekizumab. The following products will be supplied by Lilly, with study-specific labels, for use in the study:

- ixekizumab Commercial Formulation (Reference; solution for injection) in 1-mL single-dose, pre-filled, disposable manual syringes
- ixekizumab Test Formulation 1 (solution for injection) in 1-mL single-dose, pre-filled, disposable manual syringes
- ixekizumab Test Formulation 2 (solution for injection) in 1-mL single-dose, pre-filled, disposable manual syringes

## 7.2. Method of Treatment Assignment

Subjects will be randomly assigned to 1 of 3 possible treatment sequences using a computer-generated allocation code.

# 7.2.1. Selection and Timing of Doses

The actual time of all injections will be recorded in the subject's electronic case report form (eCRF).

# 7.3. Blinding

Blinding will be in place for subjects and for site staff conducting injection-site assessments and injection-site bleeding/bruising assessments.

#### 7.4. Dose Modification

Dose modification is not permitted in this study.

# 7.5. Preparation/Handling/Storage/Accountability

Investigational product will be stored refrigerated at 2°C to 8°C (36°F to 46°F) in its original carton to protect from light. Investigational product should not be frozen or shaken.

Sites will be required to monitor temperature of the on-site storage conditions of the IP. The investigator or designee must confirm appropriate temperature conditions have been maintained, as communicated by the sponsor, during transit for all IP received and ensure any discrepancies are reported and resolved before use of the study treatment.

Unblinded Site Personnel will be responsible for handling and administering IP. Unblinded Site Personnel are also responsible to make sure subjects remain blinded to treatment (ie, subjects must not see the syringe before, during or after the drug administration). Blinded assessors of injection site assessments and bleeding/bruising will not have access to the IP.

Only participants enrolled in the study may receive IP or study materials, and only authorized site staff may supply IP or administer investigational product. All IP should be stored in an environmentally controlled and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.

The investigator is responsible for study treatment accountability, reconciliation, and record maintenance (such as receipt, reconciliation, and final disposition records).

## 7.6. Treatment Compliance

The IP will be administered at the clinical site, and documentation of treatment administration will occur at the site

## 7.7. Concomitant Therapy

Subjects on stable concomitant medication at the time of study entry should continue their regular, unchanged dose throughout the study. Permitted concomitant medications include oral contraceptives, hormone replacement therapy, and thyroid replacement, at the discretion of the investigator. In addition, occasional acetaminophen is acceptable at the discretion of the investigator. However, acetaminophen should not be administered on dosing days until at least 4 hours after the injection or 4 hours before the next injection. No more than 3 g of acetaminophen will be permitted in any 24-hour period. Inclusion of subjects on any other concomitant medication is contingent upon approval following consultation with the Sponsor.

Subjects will be restricted from applying any creams or lotions on the abdominal skin the morning prior to injection and for 24 hours after injection.

If the need for any additional concomitant medication arises, continuation of the subject may be at the discretion of the investigator after consultation with a Lilly Clinical Pharmacologist (CP) or Clinical Research Physician (CRP). Any medication used during the course of the study must be documented.

# 7.8. Treatment after the End of the Study

Not applicable.

## 8. Discontinuation Criteria

Subjects discontinuing from the treatment prematurely for any reason should complete AE and other follow-up procedures per Section 2 of this protocol.

Subjects discontinuing from the study prematurely for any reason must complete AE and follow-up/ED procedures per Section 2 of this protocol.

## 8.1. Discontinuation from Study Treatment

Discontinuation of the IP for abnormal liver tests **should be considered** by the investigator when a subject meets 1 of the following conditions after consultation with the Lilly designated medical monitor:

- alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN)
- ALT or AST >3 × ULN sustained for more than 2 weeks
- ALT or AST >3 × ULN and total bilirubin level (TBL) >2 × ULN or International Normalized Ratio >1.5
- ALT or AST >3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)
- alkaline phosphatase (ALP) >3 × ULN;
- ALP  $> 2.5 \times ULN$  and TBL  $> 2 \times ULN$ ;
- ALP > 2.5 × ULN with the appearance of fatigue, nausea, vomiting, right quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

In addition, subjects will be discontinued from the study drug in the following circumstances:

- Neutrophil (segmented) counts:
  - o <500 cells/μL
  - $\circ$   $\geq$ 500 and <1000 cells/ $\mu$ L (based on 2 test results; the second test performed within 1 week from knowledge of the initial result)
  - $\circ \geq 1000$  and < 1500 cells/ $\mu L$  (based on 3 test results) and an infection that is not fully resolved
- Total white blood cell count <2000 cells/µL
- Lymphocyte count <200 cells/μL
- Platelet count <50,000 cells/μL

Subjects will also be evaluated for discontinuation from study treatment if a suicide-related thought or behavior is identified at any time during the study, or if during the study a subject gives:

- a "yes" answer to Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) on the "Suicidal Ideation" portion of the C-SSRS
- a "yes" answer to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS
- a "yes" answer to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior) on the "Suicidal Behavior" portion of the C-SSRS

In addition, subjects will also be evaluated for discontinuation from study treatment if they have self-injurious behavior that would be classified as non-suicidal self-injurious behavior, or if they had a HADS depression sub-scale ≥11 at any predose visit. It is recommended that a subject be assessed by a psychiatrist or appropriately trained professional to assist the investigator in deciding whether the subject should be discontinued from the study treatment.

## 8.1.1. Discontinuation of Inadvertently Enrolled Subjects

If the sponsor or investigator identifies a subject who did not meet enrollment criteria and was inadvertently enrolled, a discussion must occur between the Lilly CP/CRP and the investigator to determine if the subject may continue in the study. If both agree it is medically appropriate to continue, the investigator must obtain documented approval from the Lilly CP/CRP to allow the inadvertently enrolled subject to continue in the study with or without continued treatment with IP.

## 8.2. Discontinuation from the Study

Subjects will be discontinued in the following circumstances:

- Enrollment in any other clinical study involving an IP or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study
- Participation in the study needs to be stopped for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice
- Investigator Decision
  - o the investigator decides that the subject should be discontinued from the study.
- Subject Decision
  - o the subject requests to be withdrawn from the study.

Subjects discontinuing from the study prematurely for any reason must complete AE and follow-up/ED procedures per Section 2 of this protocol.

# 8.3. Subjects Lost to Follow-up

A subject will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. Site personnel are expected to make

diligent attempts to contact subjects who fail to return for a scheduled visit or were otherwise unable to be followed up by the site.
## 9. Study Assessments and Procedures

Section 2 lists the Schedule of Activities, detailing the study procedures and their timing (including tolerance limits for timing).

Appendix 2 lists the laboratory tests that will be performed for this study.

Appendix 5 provides a summary of the maximum number and volume of invasive samples, for all sampling, during the study.

Unless otherwise stated in subsections below, all samples collected for specified laboratory tests will be destroyed within 60 days of receipt of confirmed test results. Certain samples may be retained for a longer period, if necessary, to comply with applicable laws, regulations, or laboratory certification standards.

## 9.1. Efficacy Assessments

Not applicable.

#### 9.2. Adverse Events

Investigators are responsible for monitoring the safety of subjects who have entered this study and for alerting Lilly or its designee to any event that seems unusual, even if this event may be considered an unanticipated benefit to the subject.

The investigator is responsible for the appropriate medical care of subjects during the study.

Investigators must document their review of each laboratory safety report.

The investigator remains responsible for following, through an appropriate health care option, AEs that are serious or otherwise medically important, considered related to the IP or the study, or that caused the subject to discontinue the IP before completing the study. The subject should be followed until the event resolves, stabilizes with appropriate diagnostic evaluation, or is reasonably explained. The frequency of follow-up evaluations of the AE is left to the discretion of the investigator.

After the informed consent form is signed, study site personnel will record, via eCRF, the occurrence and nature of each subject's preexisting conditions. Additionally, site personnel will record any change in the condition(s) and the occurrence and nature of any AEs.

The investigator will interpret and document whether or not an AE has a reasonable possibility of being related to study treatment or a study procedure, taking into account concomitant treatment or pathologies.

A "reasonable possibility" means that there is a potential cause and effect relationship between the IP and/or study procedure and the AE.

Planned surgeries should not be reported as AEs unless the underlying medical condition has worsened during the course of the study.

#### 9.2.1. Serious Adverse Events

An SAE is any AE from this study that results in 1 of the following:

- death
- initial or prolonged inpatient hospitalization
- a life-threatening experience (that is, immediate risk of dying)
- persistent or significant disability/incapacity
- congenital anomaly/birth defect
- important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above

When a condition related to the investigational device necessitates medical or surgical intervention to preclude either permanent impairment of a body function or permanent damage to a body structure, the serious outcome of "required intervention" will be assigned. Study site personnel must alert the Lilly CRP/CP, or its designee, of any SAE as soon as practically possible.

Additionally, study site personnel must alert Lilly Global Patient Safety, or its designee, of any SAE within 24 hours of investigator awareness of the event via a sponsor-approved method. If alerts are issued via telephone, they are to be immediately followed with official notification on study-specific SAE forms. This 24-hour notification requirement refers to the initial SAE information and all follow-up SAE information.

Investigators are not obligated to actively seek AEs or SAEs in subjects once they have discontinued from and/or completed the study (the subject summary eCRF has been completed). However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably possibly related to the study treatment or study participation, the investigator must promptly notify Lilly.

Pregnancy (maternal or paternal exposure to IP) does not meet the definition of an AE. However, to fulfill regulatory requirements any pregnancy should be reported following the SAE process to collect data on the outcome for both mother and fetus.

#### 9.2.1.1. Adverse Events of Special Interest

The following AEs of special interest will be used to determine the safety and tolerability of ixekizumab injections in this clinical study.

Adverse events of special interest for ixekizumab are:

- cytopenias (leukopenia, neutropenia, and thrombocytopenia)
- liver function test changes/enzyme elevations (ALT, AST, TBL, and ALP)
- infection

- ISRs
- allergic reactions/hypersensitivities
- cerebrocardiovascular events
- malignancies
- depression
- inflammatory bowel disease (Crohn's disease and ulcerative colitis)
- interstitial lung disease

If infections, ISRs, or allergic/hypersensitivity reactions are reported, sites will provide details on these events as instructed on the eCRF. Investigators will also educate subjects about the symptoms of allergic/hypersensitivity reactions and will provide instructions on dealing with those reactions. A blood sample will be collected when possible for any subject who experiences an AE of allergic/hypersensitivity reaction during the study.

Data on cerebrocardiovascular events (defined as death, myocardial infarction, stroke, hospitalization for unstable angina, hospitalization for heart failure, coronary revascularization procedure, peripheral revascularization procedure, cardiogenic shock due to myocardial infarction, resuscitated sudden death, serious arrhythmia, hospitalization for hypertension, and peripheral arterial event) will be collected and the events will be adjudicated by an external Clinical Events Committee (CEC) made up of a chair, 2 cardiologists, and a neurologist.

Data on suspected inflammatory bowel disease, as identified by events possibly indicative of ulcerative colitis and Crohn's disease, will be collected. Suspected IBD cases will be adjudicated by an external CEC composed of gastroenterologists with expertise in inflammatory bowel disease

The role of the CEC is to adjudicate defined clinical events, in a blinded, consistent, and unbiased manner throughout the course of the study. The importance of the CECs is to ensure that all events that have been reported are evaluated uniformly by a single group.

#### 9.2.1.2. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are serious events that are not listed in the IB and that the investigator reports as related to IP or procedure. Lilly has procedures that will be followed for the recording and expedited reporting of SUSARs that are consistent with global regulations and the associated detailed guidances.

## 9.2.2. Complaint Handling

Lilly collects product complaints on IPs and drug delivery systems used in clinical trials in order to ensure the safety of study participants, monitor quality, and to facilitate process and product improvements.

Subjects should be instructed to contact the investigator as soon as possible if he or she has a complaint or problem with the IP or drug delivery system so that the situation can be assessed.

The investigator or his/her designee is responsible for handling the following aspects of the product complaint process in accordance with the instructions provided for this study:

- Recording a complete description of the product complaint reported and any associated AEs using the study-specific complaint forms provided for this purpose
- Faxing the completed Product Complaint Form within 24 hours to Lilly or its designee.

If the investigator is asked to return the product for investigation, he/she will return a copy of the Product Complaint Form with the product.

#### 9.3. Treatment of Overdose

For the purposes of this study, an overdose of ixekizumab is considered any dose higher than the dose assigned through randomization. Syringes used in this study can deliver only 1 mL volume of ixekizumab

There is no specific antidote for ixekizumab. In the event of an overdose, the subject should receive appropriate supportive care and any AEs should be documented.

Refer to the Taltz Product Label.

## 9.4. Safety

Safety will be assessed throughout the course of the study at site visits and via telephone calls in between site visits.

## 9.4.1. Laboratory Tests

For each subject, laboratory tests detailed in Appendix 2 should be conducted according to the Schedule of Activities (Section 2).

## 9.4.2. Vital Signs

For each subject, vital signs measurements should be conducted according to the Schedule of Activities (Section 2).

Blood pressure and pulse rate should be measured after at least 5 minutes sitting. Additional vital signs may be assessed as clinically indicated as well as at the scheduled times.

Unscheduled orthostatic vital signs should be assessed, if possible, during any AE of dizziness or posture-induced symptoms. Additional vital signs may be measured during each study period if warranted.

## 9.4.3. Electrocardiograms

For each subject, ECGs should be collected according to the Schedule of Activities (Section 2).

Any clinically significant findings from unscheduled ECGs that result in a diagnosis and that occur after the subject receives the first dose of the IP, should be reported to Lilly, or its designee, as an AE via eCRF.

Electrocardiograms must be recorded before collecting any blood samples. Subjects must be supine for approximately 5 to 10 minutes before ECG collection and remain supine but awake during ECG collection. Electrocardiograms may be obtained at additional times, when deemed clinically necessary. All ECGs recorded should be stored at the investigational site.

Electrocardiograms will be interpreted by a qualified physician (the investigator or qualified designee) at the site as soon after the time of ECG collection as possible, and ideally while the subject is still present, to determine whether the subject meets entry criteria at the relevant visit(s) and for immediate subject management, should any clinically relevant findings be identified.

If a clinically significant finding is identified after enrollment, the investigator will determine if the subject can continue in the study. The investigator, or qualified designee, is responsible for determining if any change in subject management is needed, and must document his/her review of the ECG printed at the time of collection. Any new clinically relevant finding should be reported as an AE.

#### 9.4.4. Temperature

Body temperature will be assessed at the times indicated in the Schedule of Activities (Section 2).

#### 9.4.5. Other Tests

#### 9.4.5.1. Injection-Site Assessments

Injection-site assessments will be performed at the times indicated in the Schedule of Activities (Section 2).

If the investigator determines that any ISR is clinically significant or if a subject indicates symptoms are indicative of an ISR (unsolicited event; volunteered by subject), the event will be captured as an AE.

Induration, swelling, pruritus, and erythema/redness associated with study injection sites will be evaluated by the blinded assessor.

## 9.4.5.2. Bleeding/Bruising Assessment

All injection sites will be observed at the times indicated in the Schedule of Activities (Section 2) by the blinded assessor, and the presence of visible bleeding/bruising will be recorded on the eCRF. A bandage may be placed on the injection site after assessment.

## 9.4.5.3. Injection-Site Pain

Pain measurements will be quantified using the 100-mm VAS pain score for all subjects. The VAS is a well-validated tool (Williamson and Hoggart 2005) to assess injection-site pain; it is presented as a 100-mm line anchored by verbal descriptors, usually "no pain" and "worst imaginable pain." The subject will be asked to relate any pain at the injection site on a scale of 1 to 100 mm on the line immediately (within 1 minute) following injection and at the time points listed in the Schedule of Activities (Section 2).

#### 9.4.5.4. Columbia Suicide Severity Rating Scale

Columbia Suicide Severity Rating Scale: a scale that captures the occurrence, severity, and frequency of suicidal ideation and/or behavior during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if suicidal ideation and/or behavior occurred. Any occurrence of suicide-related thoughts and behaviors will be assessed as indicated in the Schedule of Activities (Section 2) using the C-SSRS. The C-SSRS is administered by an appropriately trained healthcare professional with at least 1 year of patient care/clinical experience.

The nonleading AE collection should occur prior to the collection of the C-SSRS. If a suicide-related event is discovered during the C-SSRS but was not captured during the nonleading AE collection, sites should not change the AE form. If an event is serious or leads to discontinuation, this is an exception where the SAE and/or AE leading to discontinuation should be included on the AE form and the process for reporting SAEs should be followed. The first time the scale is administered in this study, the C-SSRS 'Baseline – Screening' version will be used, and the findings will constitute the baseline assessment. The C-SSRS 'Since Last Visit' scale will be used for all subsequent assessments. The Lilly Self-Harm Supplement should be completed every time the C-SSRS is administered. If there are positive findings on the Self-Harm Supplement, then the Lilly Self-Harm Follow-up form will be used to collect additional information to allow for a more complete assessment of these behaviors.

#### 9.4.5.5. Hospital Anxiety Depression Scale

The HADS depression subscale is a 7-item self-assessment scale that determines the levels of depression that a subject is experiencing over the past week. The HADS depression subscale utilizes a 4-point Likert scale (e.g., 0 to 3) for each question and is intended for ages 12 to 65 years (Zigmond and Snaith 1983; White et al. 1999). The score can range from 0 to 21, with higher scores indicating greater depression (Zigmond and Snaith 1983; Snaith 2003).

## 9.4.6. Safety Monitoring

The Lilly CP or CRP/scientist will monitor safety data throughout the course of the study.

Lilly will review SAEs within time frames mandated by company procedures. The Lilly CP or CRP will periodically review trends in safety data, laboratory analytes, and AEs.

When appropriate, the Lilly CP or CRP will consult with the functionally independent Global Patient Safety therapeutic area physician or clinical research scientist.

#### 9.4.6.1. Hepatic Safety

If a study subject experiences elevated ALT  $\geq$ 3 × ULN, ALP  $\geq$ 2 × ULN, or elevated TBL  $\geq$ 2 × ULN, liver tests (Appendix 4) should be repeated within 3 to 5 days including ALT, AST, ALP, TBL, conjugated bilirubin, gamma-glutamyl transferase, and creatinine phosphokinase to confirm the abnormality and to determine if it is increasing or decreasing. If the abnormality persists or worsens, clinical and laboratory monitoring should be initiated by the investigator based on consultation with the Lilly CP or CRP. Monitoring should continue until levels normalize and/or are returning to approximate baseline levels.

Additional safety data should be collected if 1 or more of the following conditions occur:

- elevation of serum ALT to  $\geq 5 \times ULN$  on 2 or more consecutive blood tests
- elevated serum TBL to  $\ge 2 \times \text{ULN}$  (except for cases of known Gilbert's syndrome)
- elevation of serum ALP to  $\ge 2 \times ULN$  on 2 or more consecutive blood tests
- subject discontinued from treatment due to a hepatic event or abnormality of liver tests
- hepatic event considered to be an SAE

#### 9.5. Pharmacokinetics

At the times specified in the Schedule of Activities (Section 2), venous blood samples of approximately 3 mL each will be collected. PK samples will not be analyzed for ixekizumab serum concentration unless ADA samples are also analyzed due to hypersensitivity or other adverse events, as described in Section 9.6.1.

Samples will be retained for a maximum of 1 year after the last subject visit.

## 9.6. Pharmacodynamics

Not applicable.

#### 9.6.1. Immunogenicity Assessments

At the visits and times specified in the Schedule of Activities (Section 2), venous blood samples of approximately 10 mL each will be collected to determine antibody production against ixekizumab. Due to the crossover design ADA samples will be collected and not analyzed unless clinically suggested by hypersensitivity or other AEs.

In the event of drug hypersensitivity reactions (immediate or non-immediate), additional samples will be collected as close to the onset of the event as possible, at the resolution of the event, and at least 30 days following the event. Instructions for the collection and handling of blood samples will be provided by the sponsor. The actual date and time (24-hour clock time) of each sampling will be recorded.

Samples will be retained for a maximum of 15 years after the last subject visit, or for a shorter period if local regulations and ERBs allow, at a facility selected by the sponsor. The duration allows the sponsor to respond to future regulatory requests related to ixekizumab. Any samples remaining after 15 years will be destroyed.

#### 9.7. Genetics

A blood sample will be collected for pharmacogenetic analysis as specified in the Schedule of Activities, where local regulations allow.

Samples will not be used to conduct unspecified disease or population genetic research either now or in the future. Samples will be used to investigate variable exposure or response to

ixekizumab and to investigate genetic variants thought to play a role in Ps. Assessment of variable response may include evaluation of AEs or differences in efficacy.

All samples will be coded with the subject number. These samples and any data generated can be linked back to the subject only by the investigative site personnel.

Samples will be retained for a maximum of 15 years after the last subject visit, or for a shorter period if local regulations and/or ERBs impose shorter time limits, for the study at a facility selected by Lilly or its designee. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in the development of ixekizumab.

Molecular technologies are expected to improve during the 15 year storage period and therefore cannot be specifically named. However, existing approaches include whole genome or exome sequencing, genome wide association studies, multiplex assays, and candidate gene studies. Regardless of technology utilized, data generated will be used only for the specific research scope described in this section.

#### 9.8. Biomarkers

Not applicable.

#### 9.9. Health Economics

Not applicable.

## 10. Statistical Considerations and Data Analysis

#### 10.1. Sample Size Determination

Up to 102 subjects may be enrolled to maximize the intent to have 78 subjects (26 subjects per treatment sequence) complete the study.

The objective of this study is to evaluate the injection pain immediately following dosing. Because of the crossover study design, each subject will have the opportunity to receive each treatment.

Subjects who are randomized but not administered treatment may be replaced to ensure that approximately 78 subjects may complete the study.

## 10.2. Populations for Analyses

## 10.2.1. Study Participant Disposition

A detailed description of subject disposition will be provided at the end of the study.

## 10.2.2. Study Participant Characteristics

The subjects' age, sex, weight, height, BMI, race, and other demographic characteristics will be recorded and summarized using descriptive statistics.

## 10.3. Statistical Analyses

Statistical analysis of this study will be the responsibility of Eli Lilly and Company or its designee.

Safety analyses will be conducted for all enrolled subjects who receive at least 1 dose of study drug, whether or not they completed all protocol requirements.

Continuous data will be summarized in terms of the mean, standard deviation, minimum, maximum, median, and number of observations. Categorical data will be summarized as frequency counts and percentages.

Any change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the clinical study report. Additional exploratory analyses of the data will be conducted as deemed appropriate. Complete details of the planned analyses will be documented in the Statistical Analysis Plan.

## 10.3.1. Safety Analyses

#### 10.3.1.1. Clinical Evaluation of Safety

All IP and protocol procedure AEs will be listed, and if the frequency of events allows, safety data will be summarized.

The incidence of symptoms for each treatment will be presented by severity and by association with IP as perceived by the investigator. Symptoms reported to occur prior to study entry will be distinguished from those reported as new or increased in severity during the study. Each symptom will be classified by the most suitable term from the medical regulatory dictionary.

The number of SAEs will be reported.

#### 10.3.1.2. Statistical Evaluation of Safety

#### 10.3.1.2.1. Injection-Site Pain

VAS pain score will be summarized using standard descriptive statistics. In addition, the severity of pain will be categorized by VAS pain score as: mild pain ( $\leq$ 30), moderate pain ( $\geq$ 30 and  $\leq$ 70), and severe pain ( $\geq$ 70). The number and percentage of the subjects in each pain severity category will be summarized by treatment and time point.

A mixed-effects repeated measures analysis model will be used to analyze the continuous injection-site pain VAS score by each time post-injection (0, 10, 20, 30, and 60 minutes). For measures at each time post-injection, the model will include treatment, period (Day 1, Day 8, or Day 15), treatment sequence, and treatment by treatment sequence as fixed effects. The covariance structure of the model will be unstructured. The Kenward-Roger method will be used to estimate the denominator degrees of freedom. Type III sums of squares for the least squares means will be used for the statistical comparison; treatment differences on every time point will be reported, along with the corresponding 95% confidence intervals for the differences. All pair-wise treatment comparisons by measuring time point will be evaluated and presented.

#### 10.3.1.2.2. Statistical Evaluation of Other Safety Parameters

Abnormal lab values will be listed. Other safety parameters that will be assessed include injection-site assessments, including pain, induration, swelling, pruritus, bleeding/bruising, and erythema/redness. The parameters will be listed and summarized using standard descriptive statistics. Suicidal ideation and/or behavior and self-injurious behavior with no suicidal intent, based on the C-SSRS, will be listed by subject. Only subjects that show suicidal ideation/behavior or self-injurious behavior without suicidal intent will be included in the listing (ie, if a subject answers are all 'no' for the C-SSRS, then that subject will not be displayed). HADS item scores will be listed for subjects with HADS depression sub-scale ≥11 at any time. Additional analyses may be performed if warranted upon review of the data.

## 10.3.2. Data Review During the Study

Data will be reviewed by the investigator and Sponsor throughout the course of the study to ensure subject safety.

# 10.3.3. Interim Analyses

One formal interim analysis is planned for this study. The interim analysis will include review of all available subjects' safety data (AEs, VAS, and ISR data) collected up to and including Day 21.

## 11. References

Laursen T, Hansen B, Fisker S. Pain perception after subcutaneous injections of media containing different buffers. *Basic Clin Pharmacol Toxicol*. 2006;98(2):218-221.

Snaith RP. The Hospital Anxiety and Depression Scale. *Health and Quality of Life Outcomes*. 2003;1:29. Available at: http://www.hqlo.com/content/1/1/29. Accessed October, 2018.

White D, Leach C, Sims R, Atkinson M, Cottrell D. Validation of the Hospital Anxiety and Depression Scale for use with adolescents. *Br J Psychiatry*. 1999;175(5):452-454.

Williamson A and Hoggart B. Pain: A review of three commonly used pain rating scales. *J Clin Nurs*. 2005;14(7):798-804.

Zigmond AS, Snaith RP. The Hospital Anxiety and Depression Scale. *Acta Psychiatr Scand*. 1983;67:361-370.

# Appendix 1. Abbreviations and Definitions

| Term | Definition |
|---|---|
| AE | adverse event: Any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. |
| ADA | antidrug antibodies |
| Al | autoinjector |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| BCG | Bacillus Calmette-Guérin |
| ВМІ | body mass index |
| CEC | Clinical Events Committee |
| CIOMS | Council for International Organizations of Medical Sciences |
| complaint | A complaint is any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, purity, durability, reliability, safety or effectiveness, or performance of a drug or drug delivery system. |
| compliance | Adherence to all the study-related requirements, good clinical practice requirements, and the applicable regulatory requirements. |
| confirmation | A process used to confirm that laboratory test results meet the quality requirements defined by the laboratory generating the data and that Lilly is confident that results are accurate. Confirmation will either occur immediately after initial testing or will require that samples be held to be retested at some defined time point, depending on the steps required to obtain confirmed results. |
| СР | Clinical Pharmacologist |
| CRP | Clinical Research Physician: Individual responsible for the medical conduct of the study. Responsibilities of the CRP may be performed by a physician, clinical research scientist, global safety physician or other medical officer. |
| CRU | clinical research unit |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| ECG | electrocardiogram |
| eCRF | electronic case report form |

enroll The act of assigning a subject to a treatment. Subjects who are enrolled in the study are

those who have been assigned to a treatment.

Subjects entered into a study are those who sign the informed consent form directly or enter

through their legally acceptable representatives.

**ERB** ethical review board

**GCP** good clinical practice

**HADS** Hospital Anxiety and Depression Scale

HIV human immunodeficiency virus

ΙB Investigator's Brochure

**IBD** inflammatory bowel disease

**ICF** informed consent form

**ICH** International Council for Harmonisation

lg immunoglobulin

IL interleukin

IND Investigational New Drug: An application to the FDA to allow testing of a new drug in

humans.

informed consent A process by which a subject voluntarily confirms his or her willingness to participate in a

> particular study, after having been informed of all aspects of the study that are relevant to the subject's decision to participate. Informed consent is documented by means of a

written, signed and dated informed consent form.

interim analysis An interim analysis is an analysis of clinical study data, separated into treatment groups,

that is conducted before the final reporting database is created/locked.

Investigational product (IP)

A pharmaceutical form of an active ingredient or placebo being tested or used as a reference

in a clinical study, including products already on the market when used or assembled (formulated or packaged) in a way different from the authorized form, or marketed products used for an unauthorized indication, or marketed products used to gain further information

about the authorized form.

investigator A person responsible for the conduct of the clinical study at a study site. If a study is

conducted by a team of individuals at a study site, the investigator is the responsible leader

of the team and may be called the principal investigator.

**ISR** injection-site reaction

IV intravenous

Legal

An individual or judicial or other body authorized under applicable law to consent, on Representative behalf of a prospective subject, to the subject's participation in the clinical study.

MTD maximum tolerated dose

**PFS** prefilled syringe

**Ps** psoriasis

**Q2W** every 2 weeks

**Q4W** every 4 weeks

randomize the process of assigning subjects to an experimental group on a random basis

**RBC** red blood cell

**SAE** serious adverse event

SC Subcutaneous(ly)

**screen** The act of determining if an individual meets minimum requirements to become part of a

pool of potential candidates for participation in a clinical study.

**SUSARs** suspected unexpected serious adverse reactions

**TB** tuberculosis

TBL total bilirubin level

**TEAE** treatment-emergent adverse event: Any untoward medical occurrence that emerges during

a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, and does not necessarily have to have a causal relationship with this

treatment

**TST** tuberculosis skin test

**ULN** upper limit of normal

**VAS** visual analogue scale

**WBC** white blood cell

# **Appendix 2.** Clinical Laboratory Tests

#### **Safety Laboratory Tests**

Hematology

Hematocrit Hemoglobin

Erythrocyte count (RBC) Mean cell volume Mean cell hemoglobin

Mean cell hemoglobin concentration

Leukocytes (WBC)

**Platelets** 

Differential WBC absolute counts of:

Neutrophils Lymphocytes Monocytes Eosinophils

Basophils

Urinalysis

Specific gravity

рН

Protein

Glucose Ketones

Bilirubin Urobilinogen

Blood

Nitrite
Microscopy (if dipstick abnormal)

c l

Serology

Hepatitis B surface antigen<sup>a</sup> Hepatitis B core antibody<sup>a</sup> Hepatitis C antibody<sup>a</sup>

HIV<sup>a</sup>

**Clinical Chemistry** 

Sodium Potassium Bicarbonate Chloride Calcium

Glucose (random)

Blood urea nitrogen (BUN)

Uric acid

Total cholesterol
Total protein
Albumin
Total bilirubin
Direct bilirubin
Triglycerides

Alkaline phosphatase (ALP) Aspartate aminotransferase (AST) Alanine aminotransferase (ALT)

Creatinine

Phosphorus

Other tests

Pregnancy test (females only, if applicable)<sup>b</sup>

FSH (females only, if applicable)<sup>a, c</sup> QuantiFERON $^{\mathbb{R}}$ -TB Gold or TST $^{a}$ 

Ethanol testing<sup>d</sup> Urine drug screen<sup>d</sup>

Abbreviations: FSH = follicle-stimulating hormone; HIV = human immunodeficiency virus; RBC = red blood cells; TST = tuberculin skin test; WBC = white blood cells.

- a Performed at screening only
- b Serum pregnancy test to be performed at screening. Urine pregnancy test to be performed at all other times.
- c FSH test performed for women  $\geq$ 50 and  $\leq$ 55 years of age who have had spontaneous amenhorrhea for  $\geq$ 6 months but  $\leq$ 1 year to confirm non-childbearing potential ( $\geq$ 40 mIU/mL).

d Urine drug screen and ethanol level will be performed locally at screening and at admission to the clinical research unit. Test may be repeated at additional time points at the discretion of the investigator.

# Appendix 3. Study Governance, Regulatory and Ethical Considerations

#### **Informed Consent**

The investigator is responsible for:

- ensuring that the subject understands the nature of the study, the potential risks and benefits of participating in the study, and that their participation is voluntary.
- ensuring that informed consent is given by each subject or legal representative. This includes obtaining the appropriate signatures and dates on the informed consent form (ICF) prior to the performance of any protocol procedures and prior to the administration of investigational product.
- answering any questions the subject may have throughout the study and sharing in a timely manner any new information that may be relevant to the subject's willingness to continue his or her participation in the study.
- providing a copy of the ICF to the participant or the participant's legal representative and retaining a copy on file.

#### Recruitment

Lilly or its designee is responsible for the central recruitment strategy for subjects. Individual investigators may have additional local requirements or processes. Study specific recruitment material should be approved by Lilly.

#### Ethical Review

The investigator or appropriate local representative must give assurance that the ethical review board (ERB) was properly constituted and convened as required by International Council for Harmonisation (ICH) guidelines and other applicable laws and regulations.

Documentation of ERB approval of the protocol and the ICF must be provided to Lilly before the study may begin at the investigative site(s). Lilly or its representatives must approve the ICF before it is used at the investigative site(s). All ICFs must be compliant with the ICH guideline on good clinical practice.

The study site's ERB(s) should be provided with the following:

- the current IB and Summary of Product Characteristics and updates during the course of the study
- ICF
- relevant curricula vitae

#### Regulatory Considerations

This study will be conducted in accordance with the protocol and with:

- consensus ethics principles derived from international ethics guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines
- 2) applicable ICH GCP Guidelines
- 3) applicable laws and regulations

Some of the obligations of the sponsor will be assigned to a third party organization.

## **Protocol Signatures**

The sponsor's responsible medical officer will approve the protocol, confirming that, to the best of his or her knowledge, the protocol accurately describes the planned design and conduct of the study.

After reading the protocol, each principal investigator will sign the protocol signature page and send a copy of the signed page to a Lilly representative.

## Final Report Signature

The lead investigator or designee will sign the clinical study report for this study, indicating agreement with the analyses, results, and conclusions of the report.

The sponsor's responsible medical officer and statistician will sign/approve the final clinical study report for this study, confirming that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

## Data Quality Assurance

To ensure accurate, complete, and reliable data, Lilly or its representatives will do the following:

- provide instructional material to the study sites, as appropriate.
- provide training to instruct the investigators and study coordinators. This training will give instruction on the protocol, the completion of the eCRFs, and study procedures.
- make periodic visits to the study site.
- be available for consultation and stay in contact with the study site personnel by mail, telephone, and/or fax.
- review and evaluate eCRF data and/or use standard computer edits to detect errors in data collection.
- conduct a quality review of the database.

In addition, Lilly or its representatives will periodically check a sample of the subject data recorded against source documents at the study site. The study may be audited by Lilly and/or regulatory agencies at any time. Investigators will be given notice before an audit occurs.

The investigator will keep records of all original source data. This might include laboratory tests, medical records, and clinical notes. If requested, the investigator will provide the sponsor, applicable regulatory agencies, and applicable ERBs with direct access to the original source documents.

#### Data Collection Tools/Source Data

An electronic data capture system will be used in this study. The site must define and retain all source records and must maintain a record of any data where source data are directly entered into the data capture system.

#### **Data Protection**

Data systems used for the study will have controls and requirements in accordance with local data protection law.

The purpose and use of subject personal information collected will be provided in a written document to the subject by the sponsor.

## Study and Site Closure

## **Discontinuation of Study Sites**

Study site participation may be discontinued if Lilly or its designee, the investigator, or the ERB of the study site judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

## Discontinuation of the Study

The study will be discontinued if Lilly or its designee judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice.

# Appendix 4. Hepatic Monitoring Tests for Treatment-Emergent Abnormality

Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow-up with subjects in consultation with Lilly or its designee CRP.

| Henatic | Mon | itaring | Tests |
|---------|-------|---------|--------|
| HUDAUU | TATOR | ուսլուջ | 1 6313 |

| Hepatic Hematologya | Haptoglobin <sup>a</sup> |
|---|---|
| Hemoglobin | |
| Hematocrit | Hepatic Coagulation <sup>a</sup> |
| RBC | Prothrombin Time |
| WBC | Prothrombin Time, INR |
| Neutrophils | |
| Lymphocytes | Hepatic Serologies <sup>a,b</sup> |
| Monocytes | Hepatitis A antibody, total |
| Eosinophils | Hepatitis A antibody, IgM |
| Basophils | Hepatitis B surface antigen |
| Platelets | Hepatitis B surface antibody |
| | Hepatitis B Core antibody |
| Hepatic Chemistrya | Hepatitis C antibody |
| Total bilirubin | Hepatitis E antibody, IgG |
| Conjugated bilirubin | Hepatitis E antibody, IgM |
| Alkaline phosphatase | |
| ALT | Anti-nuclear antibodya |
| AST | Alkaline Phosphatase Isoenzymesa |
| GGT | Anti-smooth muscle antibody (or anti-actin |
| СРК | antibody) <sup>a</sup> |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; CPK = creatinine phosphokinase; GGT = gamma-glutamyl transferase; Ig = immunoglobulin; INR = international normalized ratio; RBC = red blood cells; WBC = white blood cells.

- a Assayed by Lilly-designated or local laboratory.
- b Reflex/confirmation dependent on regulatory requirements and/or testing availability

# Appendix 5. Blood Sampling Summary

This table summarizes the approximate number of venipunctures and blood volumes for all blood sampling (screening, safety laboratories, and bioanalytical assays) during the study.

**Protocol I1F-MC-RHCS Sampling Summary** 

| Purpose | Blood Volume per<br>Sample (mL) <sup>b</sup> | Number of Blood<br>Samples | Total Volume (mL) <sup>b</sup> |
|---|---|---|---|
| Screening testsa | 45 / 27.7 | 1 | 45 / 27.7 |
| Clinical laboratory testsa | 12.5 / 11.7 | 6 | 75 / 70.2 |
| Pharmacokinetics | 3 | 2 | 6 |
| Immunogenicity | 10 | 3 | 30 |
| Pharmacogenetics | 10 | 1 | 10 |
| Total | | | 166 / 143.9 |
| Total for clinical purposes | | | 170 / 150 |

a Additional samples may be drawn if needed for safety purposes.

b Differing blood sample volumes pertain to different study sites.

Appendix 6. Protocol Amendment I1F-MC-RHCS (b)
Summary: A Randomized Study to Investigate
Injection-Site Pain Following Subcutaneous Injections of
2 Ixekizumab Test Formulations Compared to the
Commercial Formulation using a Pre-filled Syringe in
Healthy Subjects

#### **Overview**

Protocol I1F-MC-RHCS, A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation using a Pre-filled Syringe in Healthy Subjects, has been amended. The new protocol is indicated by Amendment (b) and will be used to conduct the study in place of any preceding version of the protocol.

Temperature assessments were added to each site visit. In addition, weekly safety telephone calls were added in between outpatient visits as appropriate.

The additional study activities were implemented to further monitor the health of subjects due to emerging data in response to a reporting of an SAE in the I1F-MC-RHCT study.

Enrollment into this study was paused in April 2019 to evaluate a potential safety concern observed in the I1F-MC-RHCT (PK Study). Approximately 80% of the VAS data had been collected; the team decided to conduct the protocol specified interim analysis based on all the available data, and stop enrolling new subjects.

## **Revised Protocol Sections**

**Note:** All deletions have been identified by strikethroughs.

All additions have been identified by the use of <u>underscore</u>.

## 1. Protocol Synopsis

Subjects may be allowed to leave the CRU after completing the 4-hour safety assessments for Day 1, at the investigator's discretion. Subjects will be readmitted to the CRU on Days 7 and 14 to receive their second and third injections on Days 8 and 15, respectively, and may be allowed to leave the CRU after completing the 4-hour safety assessments at the investigators discretion on Days 8 and 15, respectively. Subjects will return to the CRU as an outpatient on Days 21 ( $\pm 1$  day) and 43 ( $\pm 3$  days) for a safety check-up. In addition, A safety follow-up telephone calls will be conducted in between outpatient visits, on Days 28 ( $\pm 1$  day), 35 ( $\pm 3$  days), 50 ( $\pm 3$  days),  $\pm 57$  ( $\pm 3$  days), and 64 ( $\pm 3$  days), with a final safety follow-up telephone call on Day 71 ( $\pm 3$  days). There will be a follow-up visit approximately 12 weeks after the last injection.

Safety and tolerability will be assessed by monitoring of adverse events (AEs), injection-site assessments, injection-site pain, bleeding/bruising assessments, Columbia Suicide Severity Rating Scale (C-SSRS), Hospital Anxiety Depression Scale (HADS), vital signs assessments, temperature, physical examination, 12-lead electrocardiograms (ECGs), and clinical laboratory tests. Pain assessments will be made using an injection-site visual analog scale (VAS).

# 2. Schedule of Activities

| | Screening | Study Day | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -28 to -2 days<br>prior to Day<br>1 | Day<br>-1 | Day<br>1 | Day<br>7 | Day<br>8 | Day<br>14 | Day<br>15 | Day<br>21<br>(± 1<br>day) | Days<br>28 &<br>35<br>(± 3<br>days) | Day 43<br>(± 3<br>days) | Days<br>50, 57,<br>& 64<br>(± 3<br>days) | Day 71 (± 3 days) | Follow-up FU/ EDa -12 weeks post injection (±1 week) | Comments |
| Safety<br>Assessment<br>(Telephone<br>Call) | | | | | | | | | X | | X | X | (±1 week) | Every effort will be made to contact subjects as near to this time as possible but missed calls will not be recorded as protocol deviations. Subjects will be asked about the occurrence of AEs; injection-site reactions, and concomitant medication use. |
| Body<br>Temperature | | | <u>P</u> | <u>X</u> | | <u>X</u> | | <u>X</u> | | <u>X</u> | | | <u>X</u> | |

| Adverse Events and Concomitant | X | X | X | X | X | X | X | X | <u>X</u> | X | <u>X</u> | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Medication | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Follow-up / Early Discontinuation should be ~12 weeks post last injection (±1 week).

## 5. Study Design

#### 5.1 Overall Design

Subjects may be allowed to leave the CRU after completing the 4-hour safety assessments for Day 1, at the investigator's discretion. Subjects will be readmitted to the CRU on Days 7 and 14 to receive their second and third injections on Days 8 and 15, respectively, and may be allowed to leave the CRU after completing the 4-hour safety assessments at the investigators discretion on Days 8 and 15, respectively. Subjects will return to the CRU as an outpatient on Days 21 ( $\pm 1$  day) and 43 ( $\pm 3$  days) for a safety check-up. In addition, A safety follow-up telephone calls will be conducted in between outpatient visits, on Days 28 ( $\pm 1$  day), 35 ( $\pm 3$  days), 50 ( $\pm 3$  days),  $\pm 3$  days), and 64 ( $\pm 3$  days), with a final safety follow-up telephone call on Day 71 ( $\pm 3$  days). There will be a follow-up visit approximately 12 weeks after the last injection.

Safety and tolerability will be assessed by monitoring of AEs, injection-site assessments, injection-site pain, bleeding/bruising assessments, Columbia Suicide Severity Rating Scale (C-SSRS), Hospital Anxiety and Depression Scale (HADS), vital signs assessments, temperature, physical examination, 12-lead electrocardiograms (ECGs), and clinical laboratory tests.

## 5.4 Scientific Rationale for Study Design

All doses will be administered by clinical site staff to reflect safety and tolerability of the device during its intended usage.

## 7.1.2. Medical Device

The investigator or his/her designee will ensure that the instructions have been followed properly; maintaining accurate records of study devices, dispensing, and collection. The used or unused PFS may be destroyed by a qualified vendor. However, a used PFS with a product complaint will need to be returned to Lilly.

## 9.2. Adverse Events

The investigator will interpret and document whether or not an AE has a reasonable possibility of being related to study treatment, study device, or a study procedure, taking into account concomitant treatment or pathologies.

A "reasonable possibility" means that there is a potential cause and effect relationship between the IP<del>, study device</del> and/or study procedure and the AE.

## 9.3. Treatment of Overdose

For the purposes of this study, an overdose of ixekizumab is considered any dose higher than the dose assigned through randomization. <u>Syringes</u> Devices used in this study can deliver only 1 mL volume of ixekizumab.

## 9.4. **Safety**

Safety will be assessed throughout the course of the study at site visits and via telephone calls in between site visits.

## 9.4.4. Temperature

Body temperature will be assessed at the times indicated in the Schedule of Activities (Section 2).

## 10.2.3. Treatment Compliance

Every attempt will be made to select subjects who have the ability to understand and comply with instructions. Noncompliant subjects may be discontinued from the study. The time and day of administration of ixekizumab injections will be recorded. Device accountability records will be maintained by the study site.

The specifications in this protocol for the timings of safety assessments are given as targets, to be achieved within reasonable limits. Modifications may be made to the time points based upon the safety information obtained. The scheduled time points may be subject to minor alterations; however, the actual time must be correctly recorded in the eCRF.

## 10.3.2. Data Review During the Study

Data will be reviewed by the investigator <u>and Sponsor</u> throughout the course of the study to ensure subject safety.

## 10.3.3. Interim Analyses

One formal interim analysis is planned for this study. The interim analysis will include review of all <u>available</u> subjects' safety data (AEs, VAS, and ISR data) collected up to and including Day 21.